CLINICAL TRIAL: NCT04697953
Title: Brolucizumab Switch and Extend Ph IIIb Study: A Canadian, Multi-center, Single-arm, Open Label Study Assessing the Efficacy and Safety of Brolucizumab 6mg in a Treat and Extend Regimen in Patients With Neovascular Age-Related Macular Degeneration (nAMD) With Prior Anti-VEGF Exposure (PEREGRINE)
Brief Title: Efficacy and Safety of Brolucizumab 6mg in a Treat and Extend Regimen in Patients With Neovascular Age-Related Macular Degeneration (nAMD) With Prior Anti-VEGF Exposure (PEREGRINE)
Acronym: PEREGRINE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated - no participants were enrolled.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258ACA03
Record Dates: First submitted 2020-11-30; First posted 2021-01-06 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: neovascular age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — brolucizumab

STUDY DESIGN:
Intervention Model Description: Study design
  This study is a 104-week, single arm, open label, Ph IIIb multicenter study in Canadian nAMD patients.
  Neovascular AMD patients will be switched from aflibercept Q6-12W to brolucizumab at the same dosing interval at baseline. At the second visit the treating physician will conduct a disease activity assessment. If patient is stable, treatment will be extended by up to two (2) weeks using a Treat and Extend regimen interval. If the patient remains stable, the extension will also occur at next visits until maximum of Q20 Weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- brolucizumab 6mg (Experimental): Open label, brolucizumab 6mg, daily dosing, Treat & Extend regimen by up to 2 week intervals. Dosing intervals as per previous therapy and treatment extension intervals
  Interventions: Drug: brolucizumab

INTERVENTIONS:
Drug: brolucizumab — Pre-filled Syringes for intravitreal injection

SUMMARY:
The purpose of this study is to assess whether switching nAMD patients from aflibercept to brolucizumab would permit extension of treatment intervals while maintaining treatment efficacy, thereby alleviating the treatment burden on patients, caregivers, healthcare professionals (HCPs), and medical institutions.

DETAILED DESCRIPTION:
This study is a 104 week, single-arm, open label, Ph IIIb multicenter study in Canadian nAMD patients who will be switched from aflibercept 2mg to brolucizumab 6mg and extended using a Treat & Extend regimen by up to 2 week intervals assessing the durability, effectiveness, and safety of brolucizumab 6mg.

During the baseline visit, patients who consent will undergo an assessment to evaluate their eligibility based on the inclusion and exclusion criteria. Patients that meet all of the inclusion criteria and none of the exclusion criteria will be eligible to participate. The study is expected to recruit 423 patients.

If both eyes are eligible as per the inclusion and exclusion criteria, the eye with worse visual acuity should be selected for the study eye, unless the investigator deems it more appropriate to select the eye with better visual acuity.

nAMD patients stable on aflibercept q6w, q8w, q10w or q12w, will be switched to brolucizumab 6mg intravitreal injections. Disease stability is characterized by no disease activity based on the disease activity assessment (DAA) criteria (defined below) and on the investigator's judgment of visual function and/or anatomic outcomes (e.g. no change in visual acuity) or any other signs of the disease (e.g. SRF, hemorrhage, leakage, etc.).

At baseline patients will be treated with brolucizumab 6mg in the study eye only and will be scheduled for the next treatment at the pre-baseline dosing interval.

At subsequent visits, the treating physician will perform a disease activity assessment (DAA) to establish treatment extension based on the following criteria:

* Decrease in BCVA of ≥ 5 letters compared to previous visit or,
* Decrease in BCVA of ≥ 3 letters and CSFT increase ≥ 75μm compared to previous visit or,
* Any intraretinal cysts (IRC) / intraretinal fluid (IRF) compared to previous visit If the treating physician determines that there is no nAMD disease activity based on visual and anatomical assessments, i.e. no change in visual acuity and other signs of disease (e.g. IRF, SRF, hemorrhage or leakage), the following treatment can be extended by up to 2 weeks. Treatment extensions can occur at each subsequent visit to a maximum of 20 weeks between treatments.

If disease activity is identified at any study visit the interval should be shortened. If the patient is on a dosing regimen of q12w or less, the dosing interval will be shortened by two (2) weeks. For patients on a regimen of greater than q12w, the dosing interval will be shortened by four (4) weeks. If the treatment interval is currently q6w and patient fails DAA, they are not forced to discontinue, and they can be reduced to a treatment interval below q6w.

If a patient fails the first attempt to extend, the patient will have two more attempts for extension during the study.

If the patient shows significant disease activity after the second attempt for extension, injection intervals will be fixed to the previous stable, disease free interval until the end of the study.

At any point during the study, the treatment interval can also be maintained, if the investigator deems that the patient will not benefit from treatment interval adjustment (e.g., DAA due to reasons other than nAMD disease activity [e.g. fibrosis, geographic atrophy, etc.]).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained personally or by a legal proxy before any assessment is performed.
* Patients who are ≥ 50 years of age
* Confirmed diagnosis of nAMD in the judgement of the investigator
* Patients currently being treated with intravitreal injections of aflibercept 2 mg on 6-12 week dosing intervals for nAMD for a period no longer than 24 months from date of diagnosis.
* Documentation of at least one attempt to extend past the current dosing interval of aflibercept 2mg and return to stable condition at the current predefined interval
* BCVA score must be ≤ 78 (20/32) and ≥24 (20/320) letters using Early Treatment Diabetic Retinopathy Study (EDTRS)-like visual acuity charts at baseline

Exclusion Criteria:

* nAMD patients with disease activity at baseline
* Concomitant conditions or ocular disorders in the study eye at baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require planned medical or surgical intervention during the first 12-month study period.
* Simultaneous participation in a study that includes administration of any investigational drug or procedure, other than brolucizumab.
* Any active intraocular or periocular infection or active intraocular inflammation, at baseline (study eye) or in the preceding 6 months
* Uncontrolled glaucoma defined as intraocular pressure > 25 mmHg on medication, or according to investigator's judgment, at baseline (study eye)
* Patient having a fellow eye with BCVA < 20/200 at baseline due to any causes (except when due to conditions that can lead to improved VA after surgery, e.g. cataract)
* Patients who have been previously treated with brolucizumab in either eye, or who are currently receiving brolucizumab treatment in the fellow eye
* Patients who have been treated with aflibercept longer than 24 months.
* Previous use of intraocular or periocular steroids within the 6-months prior to baseline (study eye)
* Macular laser photocoagulation (focal/grid) or photodynamic therapy (PDT) at any time prior to baseline and peripheral laser photocoagulation within 3 months prior to baseline (study eye)
* Intraocular surgery within 3 months prior to baseline (except cataract; study eye) Vitreoretinal surgery at any time prior to baseline (study eye)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2021-06-21 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The proportion (%) of patients switched from aflibercept 2 mg to brolucizumab 6mg that were able to successfully extend their dosing interval at week 52 without incurring disease activity after switching | 104 weeks
  To evaluate if Neovascular Age-related Macular Degeneration (nAMD) patients can extend treatment intervals after switching from 2mg aflibercept to 6mg brolucizumab, while maintaining treatment effectiveness

SECONDARY OUTCOMES:
Mean maximum interval (number of weeks) of patients at week 104 | Up to 104 weeks
  To evaluate dosing intervals and durability of brolucizumab 6mg used in a Treat and Extend regimen after switching from aflibercept 2mg
The % of patients switched from aflibercept 2 mg to brolucizumab 6mg that were able to extend their dosing interval at week 104 | up to 104 weeks
  To evaluate dosing intervals and durability of brolucizumab 6mg used in a Treat and Extend regimen after switching from aflibercept 2mg
The % of patients switched from aflibercept 2 mg to brolucizumab 6mg that were able to maintain or extend their dosing interval at week 52 and 104 | up to 104 weeks
  To evaluate dosing intervals and durability of brolucizumab 6mg used in a Treat and Extend regimen after switching from aflibercept 2mg
Mean interval (number of weeks) of patients after switch reached at any given time point at week 52 and 104 | up to 104 weeks
  To evaluate dosing intervals and durability of brolucizumab 6mg used in a Treat and Extend regimen after switching from aflibercept 2mg
Mean change in Best Corrected Visual Acuity (BCVA) Early Treatment Diabetic Retinopathy Study (EDTRS letters) from baseline to week 52, and 104 | up to 104 weeks
  To evaluate changes in visual outcomes with brolucizumab after switching from aflibercept throughout the study in comparison to baseline assessments.
The % of patients with a change in BCVA (EDTRS letters) of 5, 10, 15 letters or more from baseline to week 52, and 104 | up to 104 weeks
  To evaluate changes in visual outcomes with brolucizumab after switching from aflibercept throughout the study in comparison to baseline assessments
The % of patients with any intraretinal fluid (IRF) and/or subretinal fluid (SRF) at baseline, weeks 52, and 104 | up to 104 weeks
  To evaluate changes of anatomical outcomes with brolucizumab after switching from aflibercept throughout the study in comparison to baseline assessments.
Incidence of ocular (e.g., intraocular infection) and non-ocular adverse events, vital signs up to week 52, and 104 | up to 104 weeks
  To evaluate safety and tolerability of treat and extend brolucizumab 6mg dosing
Mean change from baseline in central subfield foveal thickness (CSFT) | at weeks 52, 104
  To evaluate changes of anatomical outcomes with brolucizumab after switching from aflibercept throughout the study in comparison to baseline assessments.
The % of patients with pigment epithelial detachment (PED) | at baseline, weeks 52, 104
  To evaluate changes of anatomical outcomes with brolucizumab after switching from aflibercept throughout the study in comparison to baseline assessments.

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/